CLINICAL TRIAL: NCT01274546
Title: A Long-term, Multicenter Follow Up Study of the Cruciate-retaining Foundation Knee System
Brief Title: Long Term Foundation Knee Study
Status: Completed | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-705
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- "In Office": These subjects will come into the office to perform the consenting process, and complete all evaluations required at the only visit in the study.
  Interventions: Device: cruciate-retaining Foundation Knee system
- "Telephone Arm": These subjects will be consented over the phone and give a verbal consent to participate. They will complete all aspects of the study over the phone except for the knee society score evaluation and the x-ray.
  Interventions: Device: cruciate-retaining Foundation Knee system

INTERVENTIONS:
Device: cruciate-retaining Foundation Knee system — subjects who received the cruciate-retaining Foundation Knee system greater than or equal to 10 years ago and still maintain the original device in their knee.

SUMMARY:
The purpose of this study is to obtain long-term (10+ yrs) clinical and patient outcomes data on patients who received the cruciate-retaining Foundation Knee system during or prior to the year 2000.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have received a cruciate-retaining Foundation Knee system during or prior to the year 2000.
* Surgery must have been a primary knee replacement.
* Subject must have received only one primary knee replacement per hospitalization
* Subject must have had a primary diagnosis of osteoarthritis of the operative knee.
* Subject is able and willing to sign the informed consent document

Exclusion Criteria:

* Subject must not have had any previous knee implants (unicondylar or total joint replacements)
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is a prisoner

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include only subjects who received the cruciate-retaining Foundation Knee System during or before the year 2000 and who voluntarily consent to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Survivorship of the Device | Single visit
  The subject meets the inclusion/exclusion of the study and has a Foundation Knee that has survived without revision to date.

SECONDARY OUTCOMES:
Knee Society Score Evaluation | Single visit
  The knee society score includes both a subjective and a function score. The subjective score includes pain, stability and range of motion. The function score includes values for walking distance and climbing stairs.
Short Form - 36 | Single Visit
  SF-36 quality of life assessment questionnaire.
Oxford Knee Score Assessment | Single visit
  Questionnaire
WOMAC Osteoarthritis Index | Single visit
  Questionnaire
Range of Motion | Single visit
  Physician measurements of the subjects range of motion on the operated knee.
Radiographic failure | Single visit
  Radiographic failure is defined as a shift in the position of the component >3mm or 3 degrees or a >2mm radiolucency completely around the prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Friedman, M.D., Principal Investigator — Charleston Orthopedic Association; Joseph A Longo III, M.D., Principal Investigator
Locations (2):
- United States (2):
  - Scottsdale, Arizona
  - Charleston Orthopaedic Assoc., Charleston, South Carolina